CLINICAL TRIAL: NCT06655792
Title: Effectiveness of an Educational Program for Destigmatization Among Primary Health Care Providers
Brief Title: Destigmatization Among Primary Health Care Providers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Nashwan Nadhim Shwani, Lecturer, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Destigmatization
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stigma of Mental Illness
Keywords: Educational Program; Knowledge; Attitudes; Destigmatization
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Standard Care (No Educational Program) Participants in this group will not receive the educational program designed to reduce stigma toward mental illness. Instead, they will continue with their usual professional development and work routines without any specific interventions related to mental health stigma reduction.
  No intervention: This group serves as a comparison group to evaluate the effectiveness of the educational program provided to Arm 1.
  Follow-up: Similar assessments of knowledge, beliefs, and attitudes towards mental illness will be conducted before and after the study period to measure any changes that may occur in the absence of the educational intervention.
- Study Group (Experimental): Educational Program on Mental Illness Stigma Reduction
  Participants in this group will receive the educational program designed to reduce stigma toward mental illness. The educational program will be delivered through a series of structured sessions that aim to improve healthcare providers' knowledge, beliefs, and attitudes towards mental illness. These sessions will focus on the following key elements:
  Increasing knowledge about mental illness: This will include education on common mental health disorders, their symptoms, and treatments.
  Addressing misconceptions: Participants will learn about myths and misconceptions surrounding mental illness, with discussions on the importance of recognizing mental health as part of overall health.
  Promoting positive attitudes: Activities and discussions will aim to foster empathy and understanding, encouraging participants to develop supportive and non-judgmental attitudes towards individuals with mental illness.
  Interventions: Other: Educational Program on Mental Illness Stigma Reduction

INTERVENTIONS:
Other: Educational Program on Mental Illness Stigma Reduction — The intervention consists of an 8-session educational program designed to reduce stigma towards mental illness among primary healthcare providers. The program includes lectures and multimedia presentations on mental health, stigma, and its effects. It engages participants in role-playing exercises to simulate the experience of stigma and improve communication skills. Group discussions allow participants to reflect on personal beliefs and attitudes, and case studies provide real-world examples of stigma and intervention strategies. The program spans four days, with two sessions per day, each lasting 50-60 minutes.
  Arms: Study Group

SUMMARY:
The goal of this randomized controlled trial is to learn if an educational program can reduce stigma toward mental illness among primary health care providers. The main questions it aims to answer are:

* Does the educational program decrease stigma toward mental illness among participants?
* How does the program improve knowledge about mental illness?
* What beliefs about mental illness do participants hold before and after the program? Researcher will compare the intervention group, who will receive the educational program, to a control group that will not receive the program to see if the educational program is effective in reducing stigma and improving knowledge.

Participants will:

Attend educational sessions designed to increase awareness and understanding of mental illness.

Complete questionnaires about their attitudes, beliefs, and knowledge regarding mental illness before and after the program.

Provide demographic information and professional background details.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of an educational program designed to reduce stigma toward mental illness among primary health care providers in Kirkuk, Iraq. Given the critical role healthcare providers play in identifying and supporting individuals with mental health issues, addressing stigma is essential for improving mental health care delivery.

Study Design: The study will utilize a randomized controlled trial (RCT) design, with participants assigned to either an intervention group that receives the educational program or a control group that does not. This design will allow for a comparison of outcomes between the two groups.

Participants: Participants will include healthcare providers working in primary health care centers, specifically from the psychosocial, health promotion, and school health units. Primary healthcare providers within those centers will be chosen through simple random sampling to ensure a representative sample of participants.

Intervention: The educational program will consist of interactive sessions that cover topics such as the nature of mental illness, its impact on individuals and families, effective communication strategies, and methods for providing empathetic care. The program will be delivered over eight sessions, including both lectures and group discussions to facilitate engagement and learning.

Outcomes: The primary outcomes will include:

Changes in stigma levels, assessed through the Opening Minds Scale for Health Care Providers (OMS-HC).

Changes in knowledge about mental health, evaluated using the Mental Health Knowledge Questionnaire (MHKQ).

Beliefs about mental illness, measured through the Beliefs toward Mental Illness scale (BMI).

Reported and intended behaviors toward individuals with mental health problems, assessed using the Reported and Intended Behaviour Scale.

Data will be collected at three time points: pre-intervention, post-intervention, and at a follow-up stage to assess the sustainability of the program's effects.

Data Analysis: Statistical analyses will be conducted to compare pre- and post-intervention results between the intervention and control groups. Changes in stigma, knowledge, and beliefs will be analyzed to determine the program's overall effectiveness.

Significance: By evaluating the impact of this educational program, the study aims to provide evidence-based recommendations for training healthcare providers in culturally sensitive mental health care practices. Ultimately, the findings could lead to improved mental health outcomes in the community by fostering a more supportive environment for individuals experiencing mental health issues.

ELIGIBILITY:
Inclusion Criteria:

* Currently holding a position in the government health sector in Kirkuk City.
* Actively engaged in delivering assistance to clients.

Exclusion Criteria:

* Not directly involved in delivering assistance to clients.
* Unwilling to participate in the educational program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Stigma Levels | Baseline pre the educational program, and at 3 months follow-up.
  The primary outcome measure is the change in stigma levels toward mental illness among healthcare providers, as assessed by the Opening Minds Scale for Health Care Providers (OMS-HC).
  Coding\ On the 15-item scale: items 2, 6, 7, 8, 14 require reverse scoring. Outcomes: Total OMS-HC 15 mean score Total scale scores could range from 15 to 75 and a lower score indicates less stigma
  Subscales:
  1. Attitudes of health care providers towards people with mental illness (5 items = 1, 9, 10, 11, 13, 15) The concepts captured in this subscale relate to general attitudes towards people with mental illness and the role of health care providers
  2. Attitudes of health care providers towards disclosure and help-seeking (4 items = 3, 4, 5, 8) The concepts captured in this subscale relate to self-disclosure of mental illness and help seeking behavior
  3. Attitudes of health care providers towards social distance (5 items = 2, 6, 7, 12, 14)
Mental Health Knowledge Questionnaire based on educational program. | Before the educational program and at 3 months post-program completion.
  This section of the questionnaire assesses the knowledge of primary health care providers about mental health topics covered in the educational program. It consists of 10 multiple-choice questions, each presented in a "best of five" format. Participants must choose the most appropriate answer from five options. The questions are designed to evaluate key concepts such as mental illness recognition, treatment modalities, stigma reduction strategies, and best practices in patient care. The goal is to measure the impact of the educational program on enhancing the participants' understanding and competence in mental health care.

SECONDARY OUTCOMES:
Change in Knowledge About Mental Illness | Baseline pre the educational program, and at 3 month follow-up.
  The secondary outcome measure is the improvement in knowledge about mental illness, measured by the Mental Health Knowledge Questionnaire (MHKQ).
  A 16-item questionnaire, the scale consists of sixteen items rated on a dichotomous response scale (yes/no). One point is given for each 'yes' response on items 1, 3, 5, 7, 8, 11, 12, 15, 16 and 1 point is given for each 'no' response on items 2, 4, 6, 9, 10, 13 and 14. The item scores are added up to a total score (range: 0-16), with higher scores indicating higher MHK.
Change in Beliefs Toward Mental Illness | Baseline pre the educational program, and at 3 months follow-up.
  The Beliefs toward Mental Illness scale (BMI) consists of 3 subscales measuring dangerousness, Social and Interpersonal skills, and incurability. BMI is a 5-point Likert scale, consists of total 21 items, and ranging from 21 to 105. The higher score indicates more favorable beliefs towards mental illnesses
Change in Reported and Intended Behavior Toward People with Mental Illness | Baseline pre the educational program, and at 3 follow-up.
  The primary outcome measure is the change in reported and intended behavior toward people with mental illness among healthcare providers, as assessed by the Reported and Intended Behaviour Scale (RIBS).
  RIBS is a 5-points Likert scale, ranging from 4 to 20 with higher score indicates more favorable intended behavior with mentally ill patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirkuk Department of Health - Primary Health Care Sectors, Kirkuk, Kirkuk Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
Currently evaluating the feasibility of sharing IPD based on ethical considerations and institutional policies.

REFERENCES:
- [Background] Younis MS, Anwer AH, Hussain HY. Stigmatising attitude and reflections towards mental illness at community setting, population-based approach, Baghdad City 2020. Int J Soc Psychiatry. 2021 Aug;67(5):461-466. doi: 10.1177/0020764020961797. Epub 2020 Oct 8. PMID 34278834
- [Background] Tyerman J, Patovirta AL, Celestini A. How Stigma and Discrimination Influences Nursing Care of Persons Diagnosed with Mental Illness: A Systematic Review. Issues Ment Health Nurs. 2021 Feb;42(2):153-163. doi: 10.1080/01612840.2020.1789788. Epub 2020 Aug 7. PMID 32762576
- [Background] Pescosolido BA, Halpern-Manners A, Luo L, Perry B. Trends in Public Stigma of Mental Illness in the US, 1996-2018. JAMA Netw Open. 2021 Dec 1;4(12):e2140202. doi: 10.1001/jamanetworkopen.2021.40202. PMID 34932103
- [Background] Mohammadzadeh M, Awang H, Mirzaei F. Mental health stigma among Middle Eastern adolescents: A protocol for a systematic review. J Psychiatr Ment Health Nurs. 2020 Dec;27(6):829-837. doi: 10.1111/jpm.12627. Epub 2020 Apr 13. PMID 32170971
- [Background] Eiroa-Orosa FJ, Lomascolo M, Tosas-Fernandez A. Efficacy of an Intervention to Reduce Stigma Beliefs and Attitudes among Primary Care and Mental Health Professionals: Two Cluster Randomised-Controlled Trials. Int J Environ Res Public Health. 2021 Jan 29;18(3):1214. doi: 10.3390/ijerph18031214. PMID 33572955